CLINICAL TRIAL: NCT04847947
Title: The Effect of Cholecalciferol on Frailty Syndrome in Pre-frail Elderly Receiving Calcium Supplementation : A Study on Handgrip Strength, Gait Speed, Vitamin D Receptor, Insulin Growth Factor-1 and Interleukin-6
Brief Title: The Effect of Cholecalciferol in Pre-frail Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Noto Dwimartutie, , SpPD-KGer, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 72/UN2.F1/ETIK/PPM.00.02/2021
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Pre-frail Elderly
Keywords: Frailty; Pre-frail; Elderly; Cholecalciferol; Handgrip strength; Gait speed; Vitamin D receptor; Insulin Growth Factor-1; Interleukin-6
MeSH Terms: conditions — Frailty | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Oral capsule Cholecalciferol 4000 IU once daily and Calcium Lactate 500 mg once daily for 12 weeks.
  Interventions: Drug: Cholecalciferol
- Control Group (Placebo Comparator): Oral capsule Placebo once daily and Calcium Lactate 500 mg once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — Oral capsule Cholecalciferol 4000 IU once daily and Calcium Lactate 500 mg once daily for 12 weeks
  Other Names: Vitamin D3; Prove D3
  Arms: Interventional group
Drug: Placebo — Oral capsule Placebo containing white rice flour in the same identical looking with active drug once daily and Calcium Lactate 500 mg once daily for 12 weeks
  Arms: Control Group

SUMMARY:
Vitamin D plays important role in musculoskeletal health and has been known to influence immune system. Inflammaging is one of risk factors that may contribute to development of frailty in elderly.

The purpose of this study is to determine the effects of cholecalciferol in pre-frail elderly receiving calcium supplementation on handgrip strength, gait speed, vitamin D receptor, IGF-1 and IL-6. Fall incidence and improvement of frailty status will also be assessed.

DETAILED DESCRIPTION:
This is a randomized double-blind placebo-controlled study in pre-frail elderly. Measurement of frailty status based on Fried frailty phenotype criteria (weight loss, weakness, exhaustion, slowness, low physical activity level) .

Subjects who fulfill eligibility criteria will be randomized into 2 groups, one group will received cholecalciferol 4000 IU once daily and the other group will received placebo once daily. Each subjects in both groups will received calcium lactate 500 mg once daily. Intervention will be held for 12 weeks.

Handgrip strength and gait speed will be assessed at baseline, every 4 weeks, and at week 12. Other outcome measures will be assessed at baseline and at week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-frail elderly
2. Capable to understand and carry-out the instruction

Exclusion Criteria:

1. Allergic to cholecalciferol, calcium, or its components
2. Hypercalcemia (total serum calcium > 10,5 mg/dL)
3. Unwilling to stop using drug contain vitamin D or vitamin D analog or calcium
4. Using steroid or NSAID routinely
5. Acute illness during inclusion period, eg. pneumonia, stroke attack, acute exacerbation of chronic obstructive pulmonary disease, asthma attack, hypertensive urgency/emergency, acute decompensated heart failure
6. Having condition that can affect measurement of handgrip strength and gait speed, eg. hemiparesis, severe pain in extremities
7. Hepatic cirrhosis, malignancy, autoimmune disease, nephrolithiasis, malabsorption syndrome (eg. chronic diarrhea) , diabetes mellitus with HbA1c > = 8% in the last 3 months, diabetes mellitus with obvious sign and symptoms of catabolic decompensation (polyphagia, polydipsia, polyuria), chronic kidney disease stage IV-V or decreased renal function with estimated glomerular filtration rate < 30 ml/minute/1,73 m2
8. Using drug that can affect vitamin D absorption, eg. bile acid sequestrants
9. Cognitive impairment (Abbreviated Mental Test score < 8)
10. Depression (Geriatric Depression Scale score > = 10)
11. Unwilling to join the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Handgrip strength | 12 weeks (evaluation every 4 weeks)
  Change from baseline in handgrip strength. Measurement: handgrip dynamometer (Jamar Hydraulic Hand Dynamometer )
Gait speed | 12 weeks (evaluation every 4 weeks)
  Change from baseline in gait speed. Measurement: 15-feet walking test

SECONDARY OUTCOMES:
Vitamin D receptor (VDR) monocyte level | 12 weeks
  Change from baseline in VDR monocyte level. Measurement : flowcytometry
Interleukine 6 (IL-6) monocyte level | 12 weeks
  Change from baseline in IL-6 monocyte level. Measurement : flowcytometry
Insulin Growth Factor-1 (IGF-1) monocyte level | 12 weeks
  Change from baseline in IGF-1 monocyte level. Measurement : flowcytometry
serum VDR level | 12 weeks
  change from baseline in serum VDR level. Measurement : ELISA
Serum IGF-1 level | 12 weeks
  change from baseline in serum IGF-1 level. Measurement : ELISA
serum IL-6 level | 12 weeks
  change from baseline in serum IL-6 level. Measurement : ELISA
Fall incidence | 12 weeks
  number of fall
Frailty status | 12 weeks
  improvement in frailty status

CONTACTS AND LOCATIONS:
Overall Officials: Noto Dwimartutie, MD, SpPD-KGer, Principal Investigator — Division of Geriatric, Department of Internal Medicine, Faculty of Medicine Universitas Indonesia, Cipto Mangunkusumo General Hospital
Locations (1):
- Cipto Mangunkusumo General Hospital, Jakarta, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Setiati S, Anugrahini, Fransiska JE, Tamin TZ, Istanti R. Combination of alfacalcidol and calcium improved handgrip strength and mobility among Indonesian older women: A randomized controlled trial. Geriatr Gerontol Int. 2018 Mar;18(3):434-440. doi: 10.1111/ggi.13201. Epub 2017 Nov 15. PMID 29143428
- [Background] Bray NW, Doherty TJ, Montero-Odasso M. The Effect of High Dose Vitamin D3 on Physical Performance in Frail Older Adults. A Feasibility Study. J Frailty Aging. 2018;7(3):155-161. doi: 10.14283/jfa.2018.18. PMID 30095145
- [Background] Meireles MS, Kamimura MA, Dalboni MA, Giffoni de Carvalho JT, Aoike DT, Cuppari L. Effect of cholecalciferol on vitamin D-regulatory proteins in monocytes and on inflammatory markers in dialysis patients: A randomized controlled trial. Clin Nutr. 2016 Dec;35(6):1251-1258. doi: 10.1016/j.clnu.2016.04.014. Epub 2016 Apr 26. PMID 27161894